CLINICAL TRIAL: NCT05233293
Title: Comparison of SpyGlass Guided RFA On The Same Stage Versus RFA After Cytobrush for Extrahepatic Cholangiocarcinoma
Brief Title: Spyglass+RFA Versus Cytobrush+RFA for Extrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Professor, First People's Hospital of Hangzhou
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-01-10
Record Dates: First submitted 2022-01-14; First posted 2022-02-10 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Extrahepatic Cholangiocarcinoma; Malignant Biliary Obstruction
Keywords: Spyglass; RFA; extrahepatic cholangiocarcinoma; ERCP
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: parallel
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SpyGlass group (Experimental): ERCP plus SpyGlass plus RFA group
  Interventions: Procedure: Spyglass + RFA
- Cytobrush Group (Active Comparator): ERCP plus Cytobrush plus RFA group
  Interventions: Procedure: Cytobrush + RFA

INTERVENTIONS:
Procedure: Spyglass + RFA — SpyGlass direct Vision guided RFA
  Arms: SpyGlass group
Procedure: Cytobrush + RFA — After Cytobrush ,taking RFA through ERCP
  Arms: Cytobrush Group

SUMMARY:
With the development of endoscopic technology, endoscopic retrograde cholangiopancreatography (ERCP) has been widely used in the diagnosis and treatment of extrahepatic cholangiocarcinoma.In patients with extrahepatic cholangiocarcinoma, cytological brushing performed concurrently with ERCP had a lower pathologically positive rate and increased the times of ERCPs, increased the risk of postoperative complications at the same time.The present study aims to compare the efficacy and safety outcomes of Spyglass+RFA Versus Cytobrush+RFA for Extrahepatic Cholangiocarcinoma.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) has been used as the primary method for the diagnosis of biliary strictures and the treatment of extrahepatic cholangiocarcinoma. However, the accurate visual diagnosis of malignant biliary strictures and assessment of the extent of a lesion are not possible by ERCP, and treatment of extrahepatic cholangiocarcinoma by ERCP procedures is sometimes difficult. In patients with extrahepatic cholangiocarcinoma, cytological brushing performed concurrently with ERCP had a lower pathologically positive rate and increased the times of ERCPs, increased the risk of postoperative complications at the same time. Spyglass enables direct visualization of the biliary tract and the sampling of suspicious lesions, together with radiofrequency ablation.Endoscopic radiofrequency ablation (RFA) is an emerging technique for the palliation of inoperable malignant biliary strictures (MBSs). In a dozen published studies, this novel approach has shown better safety and feasibility, as well as improvement in overall survival (OS). The present study aims to compare the efficacy and safety outcomes of Spyglass+RFA Versus Cytobrush+RFA for Extrahepatic Cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years ;
* Patients with high suspicion of extrahepatic cholangiocarcinoma such as unexplained bile duct stenosis or elevated CA19-9 were found according to relevant imaging studies or symptoms;
* Willing to abide by the research procedures and sign the informed consent.

Exclusion Criteria:

* Myocardial infarction within 3 months;
* Renal insufficiency (Scr>177 umol/L);
* Serious cardiovascular and cerebrovascular or respiratory diseases before surgery;
* Preoperative shock manifestations, such as hypotension ( Systolic blood pressure <90mmHg) or increased heart rate (>120 beats/min);
* Pregnancy and lactation;
* Allergic to NSAIDs; Other clinical observation trials or those who have participated in other clinical trials within 60 days;
* Cases deemed inappropriate by the investigator (such as those with clear contraindications to ERCP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Pathological positive rate | 1 month
  Malignant tumor diagnosis rate
complications | 1 month
  Incidence of Postoperative complications such as bleeding and infection

SECONDARY OUTCOMES:
Number of sessions | 1 month
  Number of ERCP and RFA procedures
Procedure Time | Intraoperative
  Time spent for each surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Yang, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weigand K, Kuchle M, Zuber-Jerger I, Muller M, Kandulski A. Diagnostic Accuracy and Therapeutic Efficacy of Digital Single-Operator Cholangioscopy for Biliary Lesions and Stenosis. Digestion. 2021;102(5):776-782. doi: 10.1159/000513713. Epub 2021 Feb 25. PMID 33631748
- [Background] Minami H, Mukai S, Sofuni A, Tsuchiya T, Ishii K, Tanaka R, Tonozuka R, Honjo M, Yamamoto K, Nagai K, Matsunami Y, Asai Y, Kurosawa T, Kojima H, Homma T, Itoi T. Clinical Outcomes of Digital Cholangioscopy-Guided Procedures for the Diagnosis of Biliary Strictures and Treatment of Difficult Bile Duct Stones: A Single-Center Large Cohort Study. J Clin Med. 2021 Apr 12;10(8):1638. doi: 10.3390/jcm10081638. PMID 33921514